CLINICAL TRIAL: NCT06993909
Title: Clinical Approaches to Stretching Intensity in Post-Operative Knee Rehabilitation
Status: Not yet recruiting | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Other Study IDs: ACU-FTR-AOA2
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Physiotherapist
Keywords: Stretching; Post-Operative; Rehabilitation; Clinical Decision-Making

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Physiotherapists: Licensed physiotherapists with at least one year of clinical experience who have worked in post-operative knee rehabilitation within the past year. Participants will complete a one-time online or in-person questionnaire regarding their clinical decision-making on stretching intensity.

SUMMARY:
This study aims to examine how physiotherapists determine stretching intensity during knee flexion exercises in post-operative rehabilitation. It will also explore professional and clinical factors influencing these decisions, with the goal of informing standardized rehabilitation protocols.

DETAILED DESCRIPTION:
This study aims to comprehensively evaluate the approaches of physiotherapists actively involved in post-operative knee rehabilitation in determining stretching intensity during knee flexion exercises. It also seeks to identify the professional and clinical factors influencing these decisions. By revealing the variations between physiotherapists' perceptions and their actual clinical practices regarding stretching intensity, the study aims to contribute to the development of standardized clinical protocols and enhance the specificity of existing rehabilitation guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Physiotherapists with at least 1 year of clinical experience
* Involved in post-operative knee rehabilitation in the past year
* Willing to participate voluntarily

Exclusion Criteria:

* Refusal to participate
* Incomplete or inconsistent questionnaire responses

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Licensed physiotherapists in Türkiye with at least one year of clinical experience who have worked with post-operative knee rehabilitation patients within the past year.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-05-26 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Stretching Intensity in Post-Operative Knee Rehabilitation | At time of questionnaire completion (single time point)
  Primary outcome includes the duration, frequency, and maximum allowable pain/discomfort levels (measured using Visual Analog Scale) of passive knee flexion stretching exercises used by physiotherapists in post-operative rehabilitation. Data will be collected through a structured questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Acıbadem University, Ataşehir, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data (IPD) collected through the questionnaire will be made available for academic and research purposes upon reasonable request. No personally identifiable information will be included in the shared dataset.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 6 months after study completion; available for up to 3 years.
Access Criteria: Data will be made available to qualified researchers for academic and scientific purposes. Requests must include a brief research proposal and be submitted to aliomer.acar@acibadem.edu.tr.